CLINICAL TRIAL: NCT01378702
Title: Safety and Immunological Effects of Iscucin Populi and Viscum Mali e Planta Tota in Healthy Volunteers
Brief Title: Safety and Immunological Effects of Two Mistletoe Preparations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Roman Huber, Dr, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: viscum-1; 2007-002166-35 (EudraCT Number)
Record Dates: First submitted 2011-06-15; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2007-05

CONDITIONS: Healthy Volunteers
Keywords: Mistletoe; Anthroposophical medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Iscucin populi strength F, G and H (Experimental): 1 ampoule two times/week subcutaneously. Week 1-4: strength F. Week 5-8: strength G. Week 9-12: strength H.
  Interventions: Drug: mistletoe preparations
- Viscum Mali e planta tota D3, D2, 2% (Experimental): 1 ampoule two times a week subcutaneously. Week 1-4: D3. Week 4-8: D2. Week 9-12: 2%.
  Interventions: Drug: mistletoe preparations
- Placebo (Placebo Comparator): 1 ampoule two times a week subcutaneously
  Interventions: Drug: mistletoe preparations

INTERVENTIONS:
Drug: mistletoe preparations — 1 ampoule (1ml) twice per week subcutaneously
  Other Names: 1. Mistletoe from the poplar tree; 2. Mistletoe from the apple tree

SUMMARY:
The objective of this clinical trial is to describe safety, tolerability and the course of parameters of the immune system during administration of different doses of two subcutaneously administered mistletoe preparations (Iscucin populi and Viscum Mali e planta tota) in healthy volunteers, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years. Healthy volunteers

Exclusion Criteria:

* Any disease except hay fever.
* Smoking.
* Drug abuse.
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | After 4 weeks treatment with each dose
  Week 4 after baseline: evaluation of Iscucin populi strength F and Viscum Mali D3, respectively, compared to placebo. Week 8 after baseline: evaluation of Iscucin populi strength G and Viscum Mali D2, respectively, compared to placebo. Week 12 after baseline: evaluation of Iscucin populi strength H and Viscum mali 2%, respectively, compared to placebo. Week 16 after baseline: final follow up

SECONDARY OUTCOMES:
Interleukin-6 | After 4 weeks treatment with each dose
  see primary outcome measure
Eosinophil counts | After 4 weeks treatment with each dose
  see primary outcome measure
Granulocyte counts | After 4 weeks treatment with each dose
  see primary outcome measure
Lymphocyte counts | After 4 weeks treatment with each dose
  see primary outcome measure
T-cell counts | After 4 weeks treatment with each dose
  see primary outcome measure
General tolerability of the treatment(excellent, good, moderate or bad) | After 4 weeks treatment with each dose
  see primary outcome measure. Toleability will be indicated by the participants on a 4-point rating scale with the items "excellent", "good", "moderate" or "bad", which will be coded by 1, 2, 3 or 4.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Huber, Dr, Principal Investigator — University Hospital Freiburg
Locations (1):
- Univerity Medical Center Freiburg, Freiburg im Breisgau, Germany, Germany

REFERENCES:
- [Derived] Huber R, Ludtke H, Wieber J, Beckmann C. Safety and effects of two mistletoe preparations on production of Interleukin-6 and other immune parameters - a placebo controlled clinical trial in healthy subjects. BMC Complement Altern Med. 2011 Nov 24;11:116. doi: 10.1186/1472-6882-11-116. PMID 22114899
- See also: Center for Complementary Medicine, University Hospital Freiburg — http://www.uni-zentrum-naturheilkunde.de